CLINICAL TRIAL: NCT04408794
Title: A Phase 2/3 Open-label, Long-Term, Safety Trial of BHV3500 (Zavegepant*) Intranasal (IN) for the Acute Treatment of Migraine
Brief Title: Long-term Safety Study of BHV-3500 (Zavegepant*) for the Acute Treatment of Migraine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHV3500-202; C5301029 (Other: Pfizer)
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Results first posted 2023-03-16 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Acute Migraine
Keywords: migraine, headache, intranasal
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zavegepant (BHV-3500) (Experimental): 10 mg intranasal (IN) up to 8 times per month, up to 1 year
  Interventions: Drug: Zavegepant (BHV-3500)

INTERVENTIONS:
Drug: Zavegepant (BHV-3500) — 10 mg IN up to 8 times per month, up to 1 year
  Other Names: Vazegepant

SUMMARY:
The purpose of this study is to evaluate the long-term safety of BHV-3500/vazegepant intranasal in the acute treatment of migraine.

* BHV-3500, formerly "vazegepant", is now referred to as "zavegepant" (za ve' je pant). The World Health Organization (WHO) International Nonproprietary Names (INN) Expert Committee revised the name to "zavegepant" which was accepted by the United States Adopted Names (USAN ) Council for use in the U.S. and is pending formal adoption by the INN for international use.

ELIGIBILITY:
Inclusion Criteria:

* 2-8 moderate to severe migraines/month within the last 3 months
* Migraine attacks present for more than 1 year with age of onset of migraines prior to 50 years of age
* Migraine attacks, on average, lasting about 4-72 hours if untreated
* Less than 15 days with headaches (migraine or non-migraine) per month in each of the 3 months prior to the screening visit
* Ability to distinguish migraine attacks from tension/cluster headaches
* Participants with contraindications for use of triptans may be included provided they meet all other study entry criteria

Exclusion Criteria:

* History of human immunodeficiency virus disease
* History of basilar or hemiplegic migraine
* Current diagnosis of major depressive disorder requiring treatment with atypical antipsychotics, schizophrenia, bipolar disorder, or borderline personality disorder
* History of nasal surgery in the 6 months preceding the screening visit
* History of gallstones or cholecystectomy
* History of gastric, or small intestinal surgery (including gastric bypass, gastric banding, gastric sleeve, gastric balloon, etcetera), or other disease or condition (for example, chronic pancreatitis, ulcerative colitis, etcetera) that causes malabsorption.
* Body mass index ≥ 33
* Hemoglobin A1c ≥6.5%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 974 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (66):
- United States (66):
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Coastal Clinical Research, LLC, An AMR Co., Mobile, Alabama
  - Tucson Neuroscience Research, Tucson, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Pharmacology Research Institute, Encino, California
  - eStudySite, La Mesa, California
  - Synergy San Diego, Lemon Grove, California
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Wr-Pri, Llc, Newport Beach, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - California Medical Clinic for Headache, Santa Monica, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - CT Clinical Research, Cromwell, Connecticut
  - Ki Health Partners, LLC dba New England Institute for Clinical Research, Stamford, Connecticut
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - Meridien Research, Tampa, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Northwest Clinical Trials Inc., Boise, Idaho
  - Community Hospital of Anderson and Madison County Inc, Anderson, Indiana
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Collective Medical Research, Prairie Village, Kansas
  - Crescent City Headache and Neurology Center, Chalmette, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - Community Clinical Research Network, Marlborough, Massachusetts
  - Boston Neuro Research Center, South Dartmouth, Massachusetts
  - Medvadis Research Corporation, Waltham, Massachusetts
  - Michigan Headache and Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Dartmouth-Hitchcock Heater Road, Lebanon, New Hampshire
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Regional Clinical Research, Endwell, New York
  - Fieve Clinical Research, Inc, New York, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Montefiore Medical Center: Headache Center, The Bronx, New York
  - Headache Wellness Center, Greensboro, North Carolina
  - PharmQuest LLC, Greensboro, North Carolina
  - Wilmington Health, PLLC, Wilmington, North Carolina
  - OK Clinical Research LLC, Edmond, Oklahoma
  - Tekton Research, Inc., Yukon, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Union, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Volunteer Research Group, Knoxville, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Red Star Research LLC, Lake Jackson, Texas
  - DM Clinical Research, Tomball, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Jordan River Family Medicine, South Jordan, Utah
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington
  - Clinical Investigation Specialist, Inc., Kenosha, Wisconsin

REFERENCES:
- [Derived] Lipton RB, Mosher L, Fountaine RJ. Patient-Reported Outcomes During the Acute Treatment of Migraine with Zavegepant Nasal Spray: Results from a 52-Week, Open-Label Study. Pain Ther. 2026 Feb;15(1):325-340. doi: 10.1007/s40122-025-00800-z. Epub 2025 Dec 11. PMID 41379282
- [Derived] Mullin K, Croop R, Mosher L, Fullerton T, Madonia J, Lipton RB. Long-term safety of zavegepant nasal spray for the acute treatment of migraine: A phase 2/3 open-label study. Cephalalgia. 2024 Aug;44(8):3331024241259456. doi: 10.1177/03331024241259456. PMID 39210835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 63 sites in the United States.
Pre-assignment Details: A total of 974 participants were enrolled for this open-label study, of which 900 participants entered the observational phase (OP) and 608 participants entered the long-term treatment (LTT) phase, of whom 603 participants received treatment with zavegepant. A total of 286 participants failed to enter the LTT phase after the OP due to failure to meet inclusion/exclusion criteria.
Groups:
- Zavegepant 10 mg: Participants self-administered zavegepant 10 mg nasal spray, taken up to 8 times per month (28 days), for up to 52 weeks. The dose was self-administered using an Aptar Unidose System (UDS) liquid spray device.
Period: Overall Study
Arm/Group | Zavegepant 10 mg
Started (Participants in the enrolled analysis set who participated in the LTT phase, that is, non-missing interactive web response system baseline visit date.) | 608
Treated/Safety Analysis Set (Participants in the enrolled analysis set who took study drug, that is, non-missing study drug start date/time.) | 603
Completed | 341 (Participants who received the study drug and completed the study.)
Not Completed | 267
Not completed — Adverse Event | 43
Not completed — Infrequent study drug usage | 43
Not completed — Lack of Efficacy | 61
Not completed — Lost to Follow-up | 33
Not completed — Non-compliance | 6
Not completed — Physician Decision | 1
Not completed — Pregnancy | 6
Not completed — Protocol Deviation | 9
Not completed — Sheehan-STS Result | 1
Not completed — Withdrawal by Subject | 57
Not completed — Terminated study prematurely due to COVID-19 - Adverse Event | 2
Not completed — Never Treated Migraine | 5

BASELINE CHARACTERISTICS:
Population: Safety analysis set included participants in the enrolled analysis set who took the study drug, that is, non-missing study drug start date/time.
Groups:
- Zavegepant 10 mg: Participants self-administered zavegepant 10 mg nasal spray, taken up to 8 times per month (28 days), for up to 52 weeks. The dose was self-administered using an Aptar UDS liquid spray device.
Arm/Group | Zavegepant 10 mg
Number analyzed (Participants) | 603
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 517
  Male | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 71
  Not Hispanic or Latino | 532
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 23
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 70
  White | 502
  More than one race | 4
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs Leading To Discontinuation
Description: An AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in participants or clinical investigation participants administered an investigational (medicinal) product that does not necessarily have a causal relationship with this treatment. An SAE was defined as any event that met any of the following criteria at any dose: death; life-threatening; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant who received study drug; other important medical events that may not have resulted in death, be life-threatening, or required hospitalization, based upon appropriate medical judgment, they may have jeopardized the participant and may have required medical or surgical intervention to prevent one of the other serious outcomes.
Time Frame: From study drug dosing up to the end of the study (up to 52 weeks)
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Zavegepant 10 mg
Number analyzed (Participants) | 603
Participants
  AEs | 460
  SAEs | 7
  AEs leading to discontinuation | 41

2. Primary Outcome: Number Of Participants With Clinically Significant Laboratory Abnormalities
Description: Clinically significant laboratory abnormalities were defined as Grades 3 to 4 laboratory test results according to numeric laboratory test criteria found in Common Technical Criteria for Adverse Events Version 5.0 (2017) if available; otherwise, according to Division of Acquired Immune Deficiency Syndrome. Table for Grading the Severity of Adult and Pediatric Adverse Events Corrected Version 2.1 (2017) for glucose, low-density lipoprotein (LDL)-cholesterol, uric acid, and urinalysis. Laboratory test groups of clinical interest included hematology, serum chemistry, and urinalysis. Participants must have had a non-missing measurement in to be included for a given parameter. Laboratory results were presented in US units.
Time Frame: From study drug dosing up to the end of the study (up to 52 weeks)
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Zavegepant 10 mg
Number analyzed (Participants) | 579
Participants
  Alanine Aminotransferase | 3
  Aspartate Aminotransferase | 5
  Albumin: number analyzed (Participants) | 563
  Albumin | 0
  Alkaline Phosphatase | 0
  Bicarbonate: number analyzed (Participants) | 563
  Bicarbonate | 0
  Biliburin | 0
  Calcium, low: number analyzed (Participants) | 563
  Calcium, low | 0
  Calcium, high: number analyzed (Participants) | 563
  Calcium, high | 0
  Cholesterol: number analyzed (Participants) | 465
  Cholesterol | 0
  Creatine Kinase (All Methods): number analyzed (Participants) | 563
  Creatine Kinase (All Methods) | 13
  Creatine Kinase: number analyzed (Participants) | 563
  Creatine Kinase | 13
  Creatinine: number analyzed (Participants) | 564
  Creatinine | 0
  Glomerular Filtration Rate, Estimated: number analyzed (Participants) | 564
  Glomerular Filtration Rate, Estimated | 0
  LDL-cholesterol: number analyzed (Participants) | 465
  LDL-cholesterol | 21
  LDL-cholesterol, fasting: number analyzed (Participants) | 178
  LDL-cholesterol, fasting | 6
  LDL-cholesterol, not fasting: number analyzed (Participants) | 337
  LDL-cholesterol, not fasting | 15
  Lactate Dehydrogenase: number analyzed (Participants) | 562
  Lactate Dehydrogenase | 0
  Potassium, low: number analyzed (Participants) | 563
  Potassium, low | 0
  Potassium, high: number analyzed (Participants) | 563
  Potassium, high | 1
  Sodium, low: number analyzed (Participants) | 563
  Sodium, low | 0
  Sodium, high: number analyzed (Participants) | 563
  Sodium, high | 0
  Triglycerides: number analyzed (Participants) | 466
  Triglycerides | 1
  Triglycerides, fasting: number analyzed (Participants) | 179
  Triglycerides, fasting | 0
  Triglycerides, not fasting: number analyzed (Participants) | 337
  Triglycerides, not fasting | 1
  Uric Acid: number analyzed (Participants) | 563
  Uric Acid | 0
  Eosinophils: number analyzed (Participants) | 563
  Eosinophils | 0
  Hemoglobin: number analyzed (Participants) | 563
  Hemoglobin | 0
  Lymphocytes, low: number analyzed (Participants) | 563
  Lymphocytes, low | 0
  Lymphocytes, high: number analyzed (Participants) | 563
  Lymphocytes, high | 0
  Neutrophils: number analyzed (Participants) | 563
  Neutrophils | 2
  Platelets: number analyzed (Participants) | 562
  Platelets | 0
  White Blood Cells: number analyzed (Participants) | 563
  White Blood Cells | 0
  Qualitative Glucose: number analyzed (Participants) | 260
  Qualitative Glucose | 0
  Qualitative Protein: number analyzed (Participants) | 260
  Qualitative Protein | 0
  Urine Erythrocytes: number analyzed (Participants) | 78
  Urine Erythrocytes | 0

ADVERSE EVENTS:
Time Frame: From study drug dosing up to the end of the study (up to 52 weeks)
Arm/Group | Zavegepant 10 mg
All-Cause Mortality (participants affected / at risk) | 0/603
Serious Adverse Events (participants affected / at risk) | 7/603
Other Adverse Events (participants affected / at risk) | 336/603
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zavegepant 10 mg (N=603)
Appendicitis (Infections and infestations) | 1
Herpes zoster meningoencephalitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Bile duct stenosis (Hepatobiliary disorders) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Multiple sclerosis (Nervous system disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zavegepant 10 mg (N=603)
Dysgeusia (Nervous system disorders) | 236
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 62
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 33
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 33
COVID-19 (Infections and infestations) | 45
Nausea (Gastrointestinal disorders) | 37
Back pain (Musculoskeletal and connective tissue disorders) | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT04408794/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT04408794/SAP_001.pdf